CLINICAL TRIAL: NCT02374112
Title: The Effects of Medium-term Creatine Supplementation in Adults With Chronic Fatigue Syndrome
Brief Title: Creatine Supplementation in Chronic Fatigue Syndrome
Acronym: CREFAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Principal Investigator, Prof. Sergej M. Ostojic, MD, PhD, Professor, Center for Health Sciences, Serbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-2103C
Record Dates: First submitted 2015-02-22; First posted 2015-02-27 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Creatine
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Creatine supplementation
  Interventions: Dietary Supplement: Creatine
- Control (Placebo Comparator): Placebo supplementation
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine — Creatine supplementation
  Arms: Experimental
Other: Placebo — Placebo supplementation
  Arms: Control

SUMMARY:
This study evaluates the effectiveness of medium-term supplementation with creatine to improve clinical outcomes in well-defined adult CFS population. Half of the participants will receive creatine while the other half will receive placebo.

DETAILED DESCRIPTION:
Chronic fatigue syndrome (CFS) is a debilitating and complex condition characterized by profound fatigue of unknown cause, which is permanent and limits the person's functional capacity, producing various degrees of disability. It seems that inadequate or impaired energy provision through cellular metabolism may contribute to the pathogenic initiation and maintenance of CFS.

A variety of dietary interventions have been used in the management of CFS, yet no therapeutic modality demonstrated overall positive results in terms of effectiveness. Previous studies have evaluated the effects of essential fatty acids, vitamins, minerals and/or enzymes, with findings that do not support the use of a broad-spectrum nutritional supplement in treating CFS-related symptoms. Considering the fact that patients with CFS have lower levels of high-energy compounds (e.g. phosphocreatine, adenosine triphosphate), effective dietary treatment of CFS should be focused on providing compounds that facilitates cellular bioenergetics. Besides other candidate agents, creatine (Cr) could be of particular interest since it occurs naturally in the human body.

Placebo-controlled, randomized, double-blind, cross-over clinical trial examining the effectiveness of Cr for the treatment of CFS will be organized according to the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* fulfilled CDC criteria for CFS

Exclusion Criteria:

* psychiatric co-morbidity
* use of dietary supplement within 4-weeks prior to the study commencing
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI) score | 3 months

SECONDARY OUTCOMES:
health-related quality of life | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sergej M Ostojic, MD, PhD, Principal Investigator — Center for Health, Exercise and Sport Sciences

REFERENCES:
- [Background] Vermeulen RC, Kurk RM, Visser FC, Sluiter W, Scholte HR. Patients with chronic fatigue syndrome performed worse than controls in a controlled repeated exercise study despite a normal oxidative phosphorylation capacity. J Transl Med. 2010 Oct 11;8:93. doi: 10.1186/1479-5876-8-93. PMID 20937116
- [Background] Hollingsworth KG, Jones DE, Taylor R, Blamire AM, Newton JL. Impaired cardiovascular response to standing in chronic fatigue syndrome. Eur J Clin Invest. 2010 Jul;40(7):608-15. doi: 10.1111/j.1365-2362.2010.02310.x. Epub 2010 May 23. PMID 20497461